CLINICAL TRIAL: NCT06577935
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Dose-Finding Study to Evaluate the Safety, Tolerability and Efficacy of AGA2118 in Postmenopausal Women With Low Bone Mineral Density
Brief Title: A Trial Evaluating Efficacy of AGA2118 in PostMenopausal Women wIth Low Bone MasS (ARTEMIS)
Acronym: ARTEMIS
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Angitia Biopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACT23-001
Record Dates: First submitted 2024-08-14; First posted 2024-08-29 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Postmenopausal Osteoporosis
Keywords: Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- AGA2118 Dose Regimen 1 (Experimental): AGA2118 selected dose
  Participants that complete the double-blind period from study start to Month 12 will continue on to a 12 month open-label period. They will be re-randomized for Months 12 to 24.
  Interventions: Drug: AGA2118
- AGA2118 Dose Regimen 2 (Experimental): AGA2118 selected dose
  Participants that complete the double-blind period from study start to Month 12 will continue on to a 12 month open-label period. They will be re-randomized for Months 12 to 24.
  Interventions: Drug: AGA2118
- AGA2118 Dose Regimen 3 (Experimental): AGA2118 selected dose
  Participants that complete the double-blind period from study start to Month 12 will continue on to a 12 month open-label period. They will be re-randomized for Months 12 to 24.
  Interventions: Drug: AGA2118
- AGA2118 Dose Regimen 4 (Experimental): AGA2118 selected dose
  Participants that complete the double-blind period from study start to Month 12 will continue on to a 12 month open-label period. They will be re-randomized for Months 12 to 24.
  Interventions: Drug: AGA2118
- AGA2118 Dose Regimen 5 (Experimental): AGA2118 selected dose
  Participants that complete the double-blind period from study start to Month 12 will continue on to a 12 month open-label period. They will be re-randomized for Months 12 to 24.
  Interventions: Drug: AGA2118
- AGA2118 Dose Regimen 6 (Experimental): AGA2118 selected dose
  Participants that complete the double-blind period from study start to Month 12 will continue on to a 12 month open-label period. They will be re-randomized for Months 12 to 24.
  Interventions: Drug: AGA2118
- Placebo Regimen (Placebo Comparator): Placebo selected dose
  Participants that complete the double-blind period from study start to Month 12 will continue on to a 12 month open-label period. They will be re-randomized for Months 12 to 24.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: AGA2118 — Subcutaneous injection
  Arms: AGA2118 Dose Regimen 1; AGA2118 Dose Regimen 2; AGA2118 Dose Regimen 3; AGA2118 Dose Regimen 4; AGA2118 Dose Regimen 5; AGA2118 Dose Regimen 6
Other: Placebo — Subcutaneous injection
  Arms: Placebo Regimen

SUMMARY:
The primary objective of this study is to determine the effect of treatment with AGA2118 versus placebo at Month 12 on lumbar spine bone mineral density (BMD) in postmenopausal women with low bone mass.

DETAILED DESCRIPTION:
This Phase 2 dose-finding study will evaluate the safety, tolerability, and efficacy of AGA2118 at a range of dosing regimens in postmenopausal women with low BMD at the lumbar spine, total hip, or femoral neck and no prior history of fragility fractures.

This study includes a 12 month blinded treatment phase where participants will be randomized 1:1:1:1:1:1:1 to receive double-blind dosing regimens of AGA2118 or placebo. At Month 12, participants who have completed the double-blind portion of the study will continue on to a 12 month open-label period where they will be re-randomized based on their prior dosing regimen to either continue their current dosing regimen, receive a new dosing regimen, or discontinue treatment and be actively surveilled throughout Months 12 to 24.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, ambulatory, postmenopausal women age ≥ 55 to ≤ 80.
* BMD T-score of ≤ -2.5 to > -3.5 at the lumbar spine, total hip, or femoral neck.

Exclusion Criteria:

* History of vertebral fracture, or fragility fracture of the wrist, humerus, proximal femur, or pelvis.
* Vitamin D deficiency.
* Known intolerance to calcium or vitamin D supplements.
* Untreated hyper- or hypothyroidism.
* Current hyper- or hypoparathyroidism.
* Elevated transaminases.
* Significantly impaired renal function.
* Current hypo- or hypercalcemia.
* Positive for HIV, hepatitis C virus, or hepatitis B surface antigen.
* Malignancy within the last 5 years.
* Diagnosis of a familial cancer syndrome or known genetic mutation that increases risk of cancer.
* Myocardial infarction or stroke within the past 12 months.
* Use of agents affecting bone metabolism.

Ages: 55 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 379 (Actual)
Dates: Start 2024-10-31 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Percent change from Baseline to Month 12 in lumbar spine bone mineral density | 12 months
  To determine the effect of treatment with AGA2118 versus placebo at Month 12 on the percent change from Baseline in bone mineral density at the lumbar spine in postmenopausal women with low bone mineral density

SECONDARY OUTCOMES:
Percent change from Baseline to Months 3 and 6 in lumbar spine, total hip, femoral neck, and one-third distal radius bone mineral density | 3 and 6 months
  To evaluate the effect of treatment with AGA2118 versus placebo at different timepoints on percent change from Baseline in bone mineral density at the lumbar spine, total hip, femoral neck, and one-third distal radius
Percent change from Baseline to Month 12 in total hip, femoral neck, and one-third distal radius bone mineral density | 12 months
  To evaluate the effect of treatment with AGA2118 versus placebo at different timepoints on percent change from Baseline in bone mineral density at the lumbar spine, total hip, femoral neck, and one-third distal radius
Percent change from Baseline to Months 1, 3, 6, 9, and 12 in P1NP and CTX-1 | 1, 3, 6, 9, and 12 months
  To evaluate the effect of treatment with AGA2118 versus placebo at different time points on percent change from Baseline in P1NP and CTX-1
Incidence of new clinical fractures (vertebral and nonvertebral) between Baseline and Month 12 | 12 months
  To evaluate the incidence of new clinical fractures (vertebral and nonvertebral) from Baseline to Month 12

OTHER OUTCOMES:
Assessment of TEAEs (collection and documentation of all adverse events occurring during the study) | Baseline to 24 months
Number of participants who develop anti-AGA2118 antibodies | Baseline to 24 months
  To assess the formation of anti-AGA2118 antibodies
Evaluation of AGA2118 observed serum concentration levels for the AGA2118 treatment groups at Week 1 post-treatment and trough levels prior to dosing | Baseline to 24 months
  To characterize the pharmacokinetic parameters of the different AGA2118 doses

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Dent-Acosta, MD, Study Director — Angitia Incorporated Limited
Locations (23):
- United States (5):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Center for Advanced Research & Education, Gainesville, Georgia
  - NM Clinical Research & Osteoporosis Center, Inc., Albuquerque, New Mexico
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Puget Sound Osteoporosis Center, Burien, Washington
- Argentina (9):
  - Centro Médico Dra Laura Maffei e Investigación Cliínica Aplicada, Buenos Aires, Argentina
  - Consultorio de Investigacion Clinica EMO SRL, Buenos Aires, Argentina
  - IDIM, Buenos Aires, Argentina
  - Investigaciones Reumatologicas y Osteologicas SRL, Buenos Aires, Argentina
  - Mautalen - Salud e Investigacion (Expertia S.A.), Buenos Aires, Argentina
  - Stat Research, Buenos Aires, Argentina
  - Instituto Médico Strusberg, Córdoba, Argentina
  - CIDIIM, Córdoba
  - Centro de Investigaciones Medicas Mar del Plata CIM, Mar del Plata
- Poland (6):
  - Futuremeds Gdynia, Gdynia
  - Krakowskie Centrum Medyczne, Krakow
  - Futuremeds Lodz, Lodz
  - Futuremeds Warszawa Centrum, Warsaw
  - Futuremeds Targowek, Warsaw
  - Futuremeds Wroclaw, Wroclaw
- Ukraine (3):
  - CE "Hospital #1" of Zhytomyr City Council, Kyiv, Ukraine
  - Medical Center Universal Clinic "Oberig" of "Kapytal" LCC, Kyiv, Ukraine
  - PSSE Medical Centre Pulse, Vinnytsia, Ukraine